CLINICAL TRIAL: NCT04807231
Title: Comparison Between Calculated Bioavailable Testosterone Level With Radio-immunoassay Result.
Acronym: TESTOBIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0044
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Testosterone; Androgens
Keywords: testosterone; androgens; men; women
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample in order to perform a bioavailable testosterone Radio-Immuno Assay
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood withdrawal — Blood withdrawal in order to perform a bioavailable testosterone RIA (Radio-Immuno Assay).

SUMMARY:
Currently, the gold standard to obtain bioavailable testosterone results is radioimmunoassay (RIA). However, this assay requires specific equipment.

Giton in 2006 proposed an optimized calculation of the Vermeulen equation, the results of which seem to be well correlated with those obtained by RIA.

The aim of this study is to determine if the bioavailable testosterone levels determined by both methods are similar in order to replace the usual RIA assay of bioavailable testosterone by this calculation.

ELIGIBILITY:
Inclusion Criteria:

* Every men and women aged between 18 and 90 can be included

Exclusion Criteria:

* insufficient sample
* sample not send for RIA

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study is a unique cohort of 270 patients, male and female, aged between 18 and 90 (included).
  These patients have been included if there were being prescribed bioavailable testosterone by their physician in routine.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Concordance between RIA and calculated testosterone level | 2 years
  Concordance between RIA and calculated testosterone level

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No